CLINICAL TRIAL: NCT02542436
Title: An Observational Study to Investigate the Real World Effectiveness of Avastin (Bevacizumab) in the Treatment of Metastatic Colorectal Cancer in the UK
Brief Title: Avastin (Bevacizumab) in the Treatment of Metastatic Colorectal Cancer in Normal Clinical Use in the UK Population
Status: Withdrawn | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29965
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cohort 1: bevacizumab: Participants with metastatic colorectal cancer between 2010-2013, who received bevacizumab (25 mg/ml concentrate for solution for infusion) with first-line chemotherapy.
  Interventions: Other: No intervention
- Cohort 2: no bevacizumab: Participants with metastatic colorectal cancer between 2005-2008, who did not receive bevacizumab with first-line chemotherapy.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study

SUMMARY:
This study will focus on participants in the United Kingdom (UK) to collect local data on the effectiveness and safety of bevacizumab (Avastin) in the treatment of metastatic colorectal cancer in normal clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with metastatic colorectal cancer (mCRC)
* Have a Performance Status (PS) of 0-2, according to the Eastern Cooperative Oncology Group (ECOG) criteria at initiation of bevacizumab treatment
* Be chemotherapy-naive at diagnosis of mCRC or have relapsed more than 12 months after receiving adjuvant chemotherapy for early stage colorectal cancer
* Have received standard fluoropyrimidine-based chemotherapy for first-line treatment of mCRC with or without bevacizumab
* Have sufficient medical records available for assessment of eligibility at the Christie Hospital National Health Service (NHS) Trust, Manchester, United Kingdom
* For Cohort 1 (post CDF funding availability): patients between 2010-2013 who received bevacizumab with first-line chemotherapy
* For Cohort 2 (pre Cancer Drugs Fund [CDF] funding availability): patients propensity matched to cohort 1 between 2005-2008 who did not receive bevacizumab with first-line chemotherapy

Exclusion Criteria:

* Subjects with metastatic colorectal cancer, who have received bevacizumab via a clinical trial
* Subjects with metastatic colorectal cancer, whose medical records are not complete enough to confirm eligibility for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09-01 (Estimated); Primary Completion 2015-12-31 (Estimated); Study Completion 2015-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of metastatic colorectal cancer diagnosis to date of death up to 3 years

SECONDARY OUTCOMES:
Response Rate (RR) | From date of metastatic colorectal cancer diagnosis to end of study up to 3 years
Progression Free Survival (PFS) | From date of metastatic colorectal cancer diagnosis to end of study up to 3 years
Percentage of Participants with Adverse Events of Special Interest | From date of metastatic colorectal cancer diagnosis to end of study up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche